CLINICAL TRIAL: NCT05069389
Title: Registry of Management Strategies for Patients With COVID-19 in Healthcare Establishments
Acronym: HOPICOV
Status: Active, not recruiting | Type: Observational
Sponsor: Centre Hospitalier Emile Roux (Other)
Collaborators: Médipôle Lyon-Villeurbanne (Other); Centre Hospitalier Memorial France Etats-Unis (Other); Centre Hospitalier de Valence (Other); Centre Hospitalier de Troyes (Other); Groupe Hospitalier La Rochelle Ré Aunis (Unknown); Centre Hospitalier William Morey - Chalon sur Saône (Other); Centre Hospitalier de Saint-Malo (Unknown); Centre Hospitalier Intercommunal de Mont de Marsan (Unknown); Centre Hospitalier Intercommunal de Poissy / Saint-Germain (Unknown); Centre Hospitalier de Dax (Unknown); Centre Hospitalier Public du Cotentin (Unknown); Centre Hospitalier Henri Duffaut - Avignon (Other); Boulogne sur Mer Hospital Center (Other); Centre Hospitalier Louis Pasteur, Chartres (Unknown); Centre Hospitalier de Montauban (Other); Centre Hospitalier de Saint-Brieuc (Other); Groupe Hospitalier Aube Marne (Unknown)
Responsible Party: Sponsor
Other Study IDs: EDS_2020_HOPICOV
Record Dates: First submitted 2021-09-30; First posted 2021-10-06 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: COVID-19 Infection
Keywords: COVID-19; medical care strategies; hospitalisation
MeSH Terms: conditions — COVID-19 | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Data collection — Some data will be collected for all patients included :
  * specific treatment administered in COVID unit
  * dosages of treatment
  * inclusion in clinical trials
  Evolution of French recommendations and the publication of scientific articles

SUMMARY:
The purpose of the study is to describe medical care strategies implemented by healthcare establishments for patients affected by COVID-19

DETAILED DESCRIPTION:
Coronavirus infection (SARS-Cov2), very contagious, is benign in the most cases but can be complicated by an acute respiratory distress syndrome, for which an invasive mechanical ventilation in resuscitation is necessary with an important mortality rate. This infection is about an important health crisis with a fast saturation of the health system.

In front of the novelty of this virus, any effective treatment has been demonstrated in humans and researches have accelerated as this pandemic continues.

First available results, in chinese population, have not demonstrated superiority of the Lopinavir/Ritonavir association versus standard care (Cao et al. 2020). In a randomized study in 62 chinese patients, Chen et al. seems to find a clinical efficacy of the Hydroxychloroquine compared to placebo. Gautret et al. has also found a decreased viral load in nasopharyngeal swabs in patients affected by COVID-19, treated by Hydroxychloroquine and by the association of Hydroxychloroquine-Azythromycine. However, these preliminary results doesn't allow to conclue on the efficacy against COVID-19.

Currently, any treatment in particular is recommanded for patients affected by COVID-19. Randomized studies on a larger scale and greater rigor at national and european level are in process to determine the efficacy of several treatments.

Pending results of these studies, healthcare establishments had to adapt and strategize to take care their patients. These strategies have rapidely evolved during this pandemy, in terms of the therapeutic clinical studies opening, the acquisition of new knowledges on COVID-19, and treatments.

Screening : All patients with a COVID-19 diagnosis who have been treated in 2020 in participant establishements will be included in the HOPICOV study.

Enrolment : On discharge from hospital, an information notice will be delivered to the patient (or at his close relative / his legal guardian) to allow him to exert his right to oppose his collection data identified as part of the treatment. Otherwise, this information might be send by letter after his discharge.

All participating centers will be encouraged to enter data as things progress to allow interim analysis and scientific communication.

ELIGIBILITY:
Inclusion Criteria:

* Any adult patient admitted to the establishment for treatment for a SARS-Cov2 infection
* Positive RT-PCR or a scanner suggestive of COVID-19 during the stay, or with a positive serology (even if carried out after the patient's discharge)
* Hospitalization > 24h
* Patients receiving any type of care, whether it is recommended standard care or off-label treatment as part of a therapeutic clinical trial or outside the scope of clinical research

Exclusion Criteria:

* Opposition to the use of data following written patient information
* Patient transferred from another hospital to continue COVID care and whose initial care data is not available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient diagnosed for COVID-19 infection and hospitalized in healthcare establishment in 2020
Sampling Method: Non-Probability Sample
Enrollment: 2071 (Estimated)
Dates: Start 2020-06-02 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Describe management strategies implemented by healthcare establishments for patients with covid-19, depending on the evolution of scientific knowledge and recommendations for specific treatments. | During the hospitalization
  The use of specific treatments or specific care in COVID unit, inclusion in clinical trials, will be combined to report the evolution of French recommendations and scientific literature around the COVID-19.

SECONDARY OUTCOMES:
Describe management strategies to take care depending on the patient | During the hospitalization
  Specific and non specific administered treatments, inclusion in clinical trials, depending on the patients' age, symptoms at admission, comorbidities (including the presence of renal failure, unbalanced diabetes or heart disorder based on laboratory criteria and ECG) will be combined to describe different management strategies to take care depending on the patient.
Compare patients' clinical course who received different management strategies | During the hospitalization
  Comparison of hospitalization time (days), time between the onset and the end of symptoms (days), passage in intensive care and patients' vital status, according to the treatments received (non-specific / standard versus the different specific treatments administered off-label within the framework of clinical trials or not) will be combined to compare the patients' clinical course who received different management strategies
Evaluate the cost of the care | During the hospitalization
  Costs of specific treatments
Evaluate the effectiveness of the care | During the hospitalization
  Hospitalization time and survival status will be combined to evaluate the effectiveness of the care

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Center Emile Roux, Le Puy-en-Velay, France

IPD SHARING:
Plan to Share IPD: No